CLINICAL TRIAL: NCT06330883
Title: Determining the Prevalence of Frailty in COVID-19 Patients Admitted to the Intensive Care Unit and Evaluating Its Relationship With Mortality.
Brief Title: Determining the Prevalence of Frailty and Evaluating Its Relationship With Mortality.
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sinan Degirmencioglu, Research Assistant, Selcuk University
Other Study IDs: 2021/507
Record Dates: First submitted 2023-05-23; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Frailty; Mortality; COVID-19
MeSH Terms: conditions — Frailty; COVID-19 | interventions — Prognosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail: Patients will be evaluated frail if the clinical frailty score is ≥5
  Interventions: Diagnostic Test: Prognosis
- non-fragile: Patients will be evaluated non-fragile if the clinical frailty score is <5.
  Interventions: Diagnostic Test: Prognosis

INTERVENTIONS:
Diagnostic Test: Prognosis — survival/mortalite

SUMMARY:
Covid-19 patients admitted to the intensive care unit of Selcuk University Hospital were included in the study. Clinical frailty score was given during admission to the intensive care unit. Demographic data, laboratory data, radiological imaging and vital signs of the patients were recorded. Treatment and patient positions were recorded during the intensive care follow-up of the patients. Mortality status of the patients 6 months after admission to the ICU was recorded.

DETAILED DESCRIPTION:
It is planned to include non-pregnant and non-traumatic patients over the age of 18, diagnosed with COVID-19, who are treated in the Intensive Care Unit of Selcuk University Hospital. The frailty status will be evaluated by using the clinical frailty scale at the admission of the patients to the intensive care unit. Evaluation from the patient himself, if the consciousness of the patients is clear; If not, it will be done near the patient. Patients will be divided into two groups using the clinical frailty scale (CFS) as frail if the score is ≥5 and non-fragile if the score is <5. Demographic information and vaccination status (how many dose and type) will be questioned, SOFA score, APACHE II score will be recorded. Routine examinations made from the patient file; thorax computed tomography (CT) imaging, laboratory values, respiratory support information, drug treatments applied, patient positions will be recorded. Thoracic CT scans severity scores for each of the five lung lobes: 0 for no involvement (0%), 1 for minimal involvement (1%-25%), 2 for mild involvement (26-50%), 3 for moderate involvement (51%) -75) and 4 advanced involvement (76-100%). The total severity score will be the sum of the scores of the five lobes. If the score is ≤10, it will be considered as mild involvement, and if the score is >10, it will be considered as severe involvement. Laboratory values; platelet and lymphocyte count, albumin, sodium, ferritin, D-dimer, crp, procalcitonin, interleukin-6 and glomerular filtration rate values, neutrophil/lymphocyte ratio, platelet/lymphocyte ratio, CRP/Albumin ratio, arterial blood gas will be recorded. Whether or not he received respiratory support; type (invasive/non-invasive positive pressure respiratory support or high-flow nasal oxygen therapy), duration will be recorded. The use and duration of vasoactive drugs administered, renal replacement therapy and its durations will be recorded. Patient positions will be recorded as supine, lateral decubitus, and prone. The length of stay in the intensive care unit and mortality of the patients will be recorded. Comparisons will be made between frail and non-fragile groups on all these evaluated parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients who over the age of 18
* Patients who diagnosed with Covid-19

Exclusion Criteria:

* Trauma patient
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include non-pregnant and non-traumatic patients over the age of 18 who are treated with the diagnosis of COVID-19 in the Intensive Care Unit of Selcuk University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 6 months
  Mortality rate in the first 6 months after inyensive care unit admission

SECONDARY OUTCOMES:
The Sequential Organ Failure Assessment Score, The Acute Physiology and Chronic Health Evaluation II Score | First 24 hours after admission intensive care unit
  The Sequential Organ Failure Assessment score can range from a minimum of 0 to a maximum of 24 scores. Increasing scores are associated with increased hospital mortality. The Acute Physiology and Chronic Health Evaluation II Score can range from a minimum of 0 to a maximum of 71 scores. İncreasing scores are associated with increased hospital mortality.
Thorax computed tomography (CT) imaging | Within 2 weeks prior to admission ICU
  Thoracic CT scans severity scores for each of the five lung lobes: 0 for no involvement (0%), 1 for minimal involvement (1%-25%), 2 for mild involvement (26-50%), 3 for moderate involvement (51%) -75) and 4 advanced involvement (76-100%). The total severity score will be the sum of the scores of the five lobes. If the score is ≤10, it will be considered as mild involvement, and if the score is >10, it will be considered as severe involvement.
Laboratory values | Routine values at admission ICU
  Platelet and lymphocyte count, albumin, sodium, ferritin, D-dimer, crp, procalcitonin, interleukin-6 and glomerular filtration rate values, neutrophil/lymphocyte ratio, platelet/lymphocyte ratio, CRP/Albumin ratio, arterial blood gas will be recorded
Respiratory support | As long as the patient stays in the intensive care unit
  Type (invasive/non-invasive positive pressure respiratory support or high-flow nasal oxygen therapy), duration will be recorded
Vasoactive drugs administered | Data will be collected from the admission to the intensive care unit up to 6 months or until mortality within this period.
  Starting from the admission of patients to the intensive care unit, vasoactive drug records will be kept daily until either the patient's mortality in the intensive care unit or their discharge from the intensive care unit, up to a maximum of 6 months from admission to the intensive care unit.
Renal replacement therapy | Data will be collected from the admission to the intensive care unit up to 6 months or until mortality within this period.
  Total time the patient used renal replacement therapy as long as he stayed in the intensive care unit
Patient positions | Data will be collected from the admission to the intensive care unit up to 6 months or until mortality within this period.
  Patient positions will be recorded as supine, lateral decubitus, and prone.
Length of stay in the intensive care unit | Data will be collected from the admission to the intensive care unit up to 6 months or until mortality within this period.
  The number of calendar days from the date of admission to the intensive care unit until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jale Bengi Çelik, Study Director — Selcuk University Hospital, Department of Anesthesiology and Reanimation, jalecelik@hotmail.com
Locations (1):
- Selcuk University Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No